CLINICAL TRIAL: NCT01136174
Title: A Double-blind, Randomised, Placebo-controlled (Within a Dose Group) Study to Evaluate Safety and Pharmacokinetics of Multiple Rising Doses of BIBF 1120 at 50 mg Bid (14 Days), 100 mg Bid (14 Days), and 150 mg Bid (28 Days) p.o., on Top of Standard Medical Care With Stratification According to Pirfenidone Use, in Japanese Patients With Idiopathic Pulmonary Fibrosis.
Brief Title: Safety and PK Study of BIBF 1120 in Japanese Patients With IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1199.31
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

ARMS (4):
- BIBF 1120 50 mg (Experimental): Low dose for cohort 1
  Interventions: Drug: BIBF 1120
- BIBF 1120 100 mg (Experimental): Middle dose for cohort 2
  Interventions: Drug: BIBF 1120
- BIBF 1120 150 mg (Experimental): High dose for cohort 3
  Interventions: Drug: BIBF 1120
- Placebo (Placebo Comparator): Placebo for cohort 1,2,3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo BID for cohort 1,2,3
  Arms: Placebo
Drug: BIBF 1120 — 50 mg, 100 mg, 150 mg BID will be used for Cohort 1, 2, and 3 respectively
  Arms: BIBF 1120 50 mg
Drug: BIBF 1120 — 50 mg, 100 mg, 150 mg BID will be used for Cohort 1, 2, and 3 respectively
  Arms: BIBF 1120 100 mg
Drug: BIBF 1120 — 50 mg, 100 mg, 150 mg BID will be used for Cohort 1, 2, and 3 respectively
  Arms: BIBF 1120 150 mg

SUMMARY:
To investigate safety of BIBF 1120 in Japanese patients with idiopathic pulmonary fibrosis (IPF), with and without pirfenidone background treatment.

To assess pharmacokinetics of BIBF 1120 in Japanese patients, with and without pirfenidone background treatment.

To assess pharmacokinetics of pirfenidone in Japanese patients, alone and in combination with BIBF 1120 treatment.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of idiopathic pulmonary fibrosis (IPF) according to American Thoracic Society (ATS) /European Respiratory Society (ERS) guideline
2. Forced vital capacity (FVC) 50-90%
3. Diffusing capacity for carbon monoxide (DLCO) 30-79%
4. For patients on pirfenidone, have been on a steady dose for at least 3 months

Exclusion criteria:

1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 1.5 x upper limit of normal range (ULN) at screening.
2. Bilirubin > 1.5 x ULN at screening.
3. Relevant airways obstruction (i.e. pre-bronchodilator FEV1/FVC <0.7) at screening.
4. Continuous oxygen supplementation.
5. Active infection at screening or randomisation.
6. Being treated with any of the following concomitant medications.

   * Oral corticosteroid medication at unstable dose
   * ketoconazole or atazanavir
7. Patients who are expected to go on to lung transplantation, have rapidly deteriorating disease, or have a life expectancy less than 3 months from screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (8):
- Japan (8):
  - 1199.31.002 Boehringer Ingelheim Investigational Site, Bunkyo-ku,Tokyo
  - 1199.31.004 Boehringer Ingelheim Investigational Site, Hamamatsu, Shizuoka
  - 1199.31.008 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1199.31.006 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1199.31.007 Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - 1199.31.005 Boehringer Ingelheim Investigational Site, Seto, Aichi
  - 1199.31.001 Boehringer Ingelheim Investigational Site, Shimotsuke,Tochigi
  - 1199.31.003 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

REFERENCES:
- [Derived] Ogura T, Taniguchi H, Azuma A, Inoue Y, Kondoh Y, Hasegawa Y, Bando M, Abe S, Mochizuki Y, Chida K, Kluglich M, Fujimoto T, Okazaki K, Tadayasu Y, Sakamoto W, Sugiyama Y. Safety and pharmacokinetics of nintedanib and pirfenidone in idiopathic pulmonary fibrosis. Eur Respir J. 2015 May;45(5):1382-92. doi: 10.1183/09031936.00198013. Epub 2014 Dec 10. PMID 25504994

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo oral administration twice a day
- BIBF 1120 50 mg: BIBF 1120 50 mg oral administration twice a day
- BIBF 1120 100 mg: BIBF 1120 100 mg oral administration twice a day
- BIBF 1120 150 mg: BIBF 1120 150 mg oral administration twice a day
Period: Overall Study
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Started | 12 | 6 | 8 | 24
Completed | 12 | 6 | 8 | 20
Not Completed | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who received study medication and were documented to have taken at least one dose of investigational treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg | Total
Number analyzed (Participants) | 12 | 6 | 8 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.3) | 66.7 (2.9) | 67.5 (7.4) | 64.7 (8.5) | 65.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 8 | 15
  Male | 11 | 4 | 4 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Drug-related Adverse Events
Description: The number of patients with drug-related adverse events stratified according to pirfenidone use in each group
Time Frame: after the first drug intake until 28 days from the last treatment administration, up to 60 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 12 | 6 | 8 | 24
participants
  Patients with Pirfenidone (N = 5, 4, 4, 13) | 1 | 0 | 0 | 7
  Patients without Pirfenidone (N = 7, 2, 4, 11) | 1 | 0 | 1 | 3

2. Secondary Outcome: AUCτ,ss After Multiple Doses of BIBF 1120 Without Pirfenidone
Description: AUCτ,ss was calculated as the area under the concentration-time curve of the concentration-time profile of the analyte in plasma at steady state over a uniform dosing interval τ after multiple doses of BIBF 1120 without pirfenidone in the time frame mentioned.
  Detailed outcome measure time frame:
  In 50 mg and 100 mg dose group:
  BIBF 1120:
  days 14 (-1, +3) to 17 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
  In 150 mg dose group:
  BIBF 1120:
  days 28 (-1, +3) to 31 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
Time Frame: pre-dose, then 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose on days 14 to 17 (BIBF 1120 50 mg and 100 mg) or on days 28 to 31 (BIBF 1120 150 mg)
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 2 | 4 | 9
ng*h/mL | 33.7 (165) | 115 (32.4) | 218 (58.3)

3. Secondary Outcome: Cmax,ss After Multiple Doses of BIBF 1120 Without Pirfenidone
Description: Maximum measured concentration of the analyte in plasma at steady state was identified from measurements obtained at multiple time points over a uniform dosing interval τ after multiple doses of BIBF 1120 without pirfenidone.
  Detailed outcome measure time frame:
  In 50 mg and 100 mg dose group:
  BIBF 1120:
  days 14 (-1, +3) to 17 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
  In 150 mg dose group:
  BIBF 1120:
  days 28 (-1, +3) to 31 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
Time Frame: as for outcome 2
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 2 | 4 | 9
ng/mL | 9.09 (173) | 20.0 (64.5) | 39.7 (68.1)

4. Secondary Outcome: AUCτ,ss After Multiple Doses of BIBF 1120 With Pirfenidone
Description: AUCτ,ss was calculated as the area under the concentration-time curve of the concentration-time profile of the analyte in plasma at steady state over a uniform dosing interval τ after multiple doses of BIBF 1120 with pirfenidone in the time frame mentioned.
  Detailed outcome measure time frame:
  In 50 mg and 100 mg dose group:
  BIBF 1120:
  days 14 (-1, +3) to 17 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
  In 150 mg dose group:
  BIBF 1120:
  days 28 (-1, +3) to 31 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
Time Frame: as for outcome 2
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 3 | 7
ng*h/mL | 67.9 (16.7) | 86.0 (62.7) | 149 (18.0)

5. Secondary Outcome: Cmax,ss After Multiple Doses of BIBF 1120 With Pirfenidone
Description: Maximum measured concentration of the analyte in plasma at steady state was identified from measurements obtained at multiple time points over a uniform dosing interval τ after multiple doses of BIBF 1120 with pirfenidone
  Detailed outcome measure time frame:
  In 50 mg and 100 mg dose group:
  BIBF 1120:
  days 14 (-1, +3) to 17 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
  In 150 mg dose group:
  BIBF 1120:
  days 28 (-1, +3) to 31 at Visit 5: At pre-dose and 0.5 h, 1 h, 2 h, 3 h, 3.92 h, 6 h, 8 h, 12 h, 24 h, 48 h, 72 h after morning dose
Time Frame: as for outcome 2
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 3 | 7
ng/mL | 10.9 (50.3) | 13.8 (113) | 23.5 (27.2)

6. Secondary Outcome: AUC0-4,ss After Multiple Doses of Pirfenidone 600 mg Without BIBF 1120 (After Breakfast)
Description: AUC0-4,ss was calculated as the area under the curve of the concentration-time profile of the analyte in plasma at steady state over the time interval from 0 to 4 hours after multiple doses of Pirfenidone 600 mg without BIBF 1120 (after breakfast) in the time frame mentioned.
Time Frame: Day -1 at Visit 1: At pre-dose and 0.5 h, 1 h, 2 h, 3 h after morning dose and pre-dose after lunch dose
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 3 | 9
ng*h/mL | 28900 (30.7) | 34400 (36.3) | 45800 (26.6) | 32500 (21.2)

7. Secondary Outcome: Cmax,ss After Multiple Doses of Pirfenidone 600 mg Without BIBF 1120 (After Breakfast)
Description: Maximum measured concentration of the analyte in plasma at steady state was identified from measurements obtained at multiple time points after multiple doses of Pirfenidone 600 mg without BIBF 1120 (after breakfast)
Time Frame: Day -1 at Visit 1: At pre-dose and 0.5 h, 1 h, 2 h, 3 h after morning dose and pre-dose after lunch dose
Population: Treated set-Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 4 | 9
ng/mL | 11300 (22.1) | 11900 (28.9) | 14600 (41.5) | 11200 (26.6)

8. Secondary Outcome: AUC0-4,ss After Multiple Doses of Pirfenidone 600 mg With BIBF 1120 (After Breakfast)
Description: AUC0-4,ss was calculated as the area under the concentration-time curve of the concentration-time profile of the analyte in plasma at steady state over the time interval from 0 to 4 hours after multiple doses of Pirfenidone 600 mg with BIBF 1120 (after breakfast) in the time frame mentioned.
Time Frame: Day 14 at Visit 5 (BIBF 1120 50mg and 100mg) and day 28 (visit 7) (BIBF 1120 150mg): At pre-dose and 0.5 h, 1 h, 2 h, 3 h after morning dose and pre-dose after lunch dose
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 3 | 7
ng*h/mL | 28800 (6.85) | 34300 (39.9) | 35000 (32.2) | 35900 (21.8)

9. Secondary Outcome: Cmax,ss After Multiple Doses of Pirfenidone 600 mg With BIBF 1120 (After Breakfast)
Description: Maximum measured concentration of the analyte in plasma at steady state was identified from measurements obtained at multiple time points after multiple doses of Pirfenidone 600 mg with BIBF 1120 (after breakfast)
Time Frame: as for outcome 8
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 3 | 8
ng/mL | 12000 (23.1) | 12800 (44.3) | 15300 (51.1) | 12600 (27.2)

10. Secondary Outcome: AUC0-8,ss After Multiple Doses of Pirfenidone 600 mg Without BIBF 1120 (After Lunch)
Description: AUC0-8,ss was calculated as the area under the concentration-time curve of the concentration-time profile of the analyte in plasma at steady state over the time interval from 0 to 8 hours after multiple doses of Pirfenidone 600 mg without BIBF 1120 (after lunch) in the time frame mentioned.
Time Frame: Day -1 at Visit 1: at pre-dose and 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h after lunch dose
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 3 | 8
ng*h/mL | 56600 (25.8) | 72800 (40.7) | 84100 (11.4) | 60900 (22.9)

11. Secondary Outcome: Cmax,ss After Multiple Doses of Pirfenidone 600 mg Without BIBF 1120 (After Lunch)
Description: Maximum measured concentration of the analyte in plasma at steady state was identified from measurements obtained at multiple time points after multiple doses of Pirfenidone 600 mg Without BIBF 1120 (after lunch)
Time Frame: Day -1 at Visit 1: at pre-dose and 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h after lunch dose
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 4 | 9
ng/mL | 13500 (19.9) | 14600 (20.9) | 15100 (19.5) | 12900 (30.2)

12. Secondary Outcome: AUC0-8,ss After Multiple Doses of Pirfenidone 600 mg With BIBF 1120 (After Lunch)
Description: AUC0-8,ss was calculated as the area under the concentration-time curve of the concentration-time profile of the analyte in plasma at steady state over the time interval from 0 to 8 hours after multiple doses of Pirfenidone 600 mg with BIBF 1120 (after lunch) in the time frame mentioned.
Time Frame: Day 14 at Visit 5 (BIBF 1120 50mg and 100mg) and day 28 (visit 7) (BIBF 1120 150mg): at pre-dose and 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h after lunch dose
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 3 | 6
ng*h/mL | 47000 (13.6) | 71000 (40.8) | 71500 (19.1) | 63600 (27.7)

13. Secondary Outcome: Cmax,ss After Multiple Doses of Pirfenidone 600 mg With BIBF 1120 (After Lunch)
Description: Maximum measured concentration of the analyte in plasma at steady state was identified from measurements obtained at multiple time points after multiple doses of Pirfenidone 600 mg with BIBF 1120 (after lunch)
Time Frame: as for outcome 12
Population: Treated set- Only patients with valid final pharmacokinetic values were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 4 | 4 | 3 | 8
ng/mL | 10700 (18.8) | 12000 (37.3) | 12100 (10.7) | 12500 (23.0)

14. Secondary Outcome: Withdrawal Due to Adverse Event
Description: Number of patients prematurely discontinued from trial medication due to adverse event.
Time Frame: after the first drug intake until 28 days from the last treatment administration, up to 60 days
Population: Treated set
Measure: Number; unit: participants
Groups:
- Placebo: Placebo oral administration twice a day for cohort 1, 2, 3
- BIBF 1120 50 mg: BIBF 1120 50 mg oral administration twice a day for cohort 1
- BIBF 1120 100 mg: BIBF 1120 100 mg oral administration twice a day for cohort 2
- BIBF 1120 150 mg: BIBF 1120 150 mg oral administration twice a day for cohort 3
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 12 | 6 | 8 | 24
participants
  With Pirfenidone (N= 5, 4, 4, 13) | 0 | 0 | 0 | 2
  Without Pirfenidone (N = 7, 2, 4, 11) | 0 | 0 | 0 | 2

15. Secondary Outcome: Clinical Relevant Abnormalities in Laboratory Parameters- No Pirfenidone Background
Description: Number of patients with Clinical Relevant Abnormalities in laboratory parameters reported as adverse events - No pirfenidone background
Time Frame: after the first drug intake until 28 days from the last treatment administration, up to 60 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 7 | 2 | 4 | 11
participants
  Alanine aminotransferase increased | 0 | 0 | 0 | 2
  Aspartate aminotransferase increased | 0 | 0 | 0 | 2
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 1
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 1

16. Secondary Outcome: Clinical Relevant Abnormalities in Laboratory Parameters- With Pirfenidone Background
Description: Number of patients with Clinical Relevant Abnormalities in laboratory parameters reported as adverse events - With pirfenidone background
Time Frame: after the first drug intake until 28 days from the last treatment administration, up to 60 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Number analyzed (Participants) | 5 | 4 | 4 | 13
participants
  Hypothyroidism | 0 | 0 | 0 | 1
  Transaminases increased | 0 | 0 | 0 | 1

17. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Placebo oral administration twice a day for cohort 3
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 24
mmHg
  DBP | 0.5 (13.3) | -0.8 (10.8)
  SBP | 1.3 (19.2) | 2.5 (14.4)

18. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline in pulse rate at day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 24
bpm | -2.5 (15.4) | 1.9 (13.6)

19. Secondary Outcome: Lung Function Measurement: Diffusing Capacity for Carbon Monoxide (DLco)
Description: Change in diffusing capacity for carbon monoxide (DLco) from baseline to day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 24
mL/min/mmHg | -1.131 (1.397) | -0.707 (2.005)

20. Secondary Outcome: Lung Function Measurement: Diffusing Capacity for Carbon Monoxide Percent of Predicted (%DLco)
Description: Change in Diffusing Capacity for Carbon Monoxide percent of predicted (%DLco) from baseline to day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set- Only patients with valid measurements were analysed.
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 23
% predicted | -4.660 (8.020) | -1.193 (5.948)

21. Secondary Outcome: Lung Function Measurement: Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in forced expiratory volume in 1 second (FEV1) from baseline to day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 24
Liter | -0.021 (0.107) | 0.036 (0.078)

22. Secondary Outcome: Lung Function Measurement: Forced Vital Capacity (FVC)
Description: Change in forced vital capacity (FVC) from baseline to day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 24
Liter | -0.081 (0.175) | 0.050 (0.086)

23. Secondary Outcome: Lung Function Measurement: Forced Vital Capacity Percent of Predicted (%FVC)
Description: Change in Forced Vital Capacity percent of predicted (%FVC) from baseline to day 35. Only the results for placebo and Nintedanib 150mg arm were reported for this endpoint as nintedanib 150mg is the target dose.
Time Frame: baseline and day 35
Population: Treated set
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Placebo | BIBF 1120 150 mg
Number analyzed (Participants) | 8 | 24
% predicted | -2.311 (5.193) | 1.432 (2.671)

ADVERSE EVENTS:
Time Frame: after the first drug intake until 28 days from the last treatment administration, up to 60 days
Arm/Group | Placebo | BIBF 1120 50 mg | BIBF 1120 100 mg | BIBF 1120 150 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/8 | 1/24
Other Adverse Events (participants affected / at risk) | 4/12 | 0/6 | 4/8 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | BIBF 1120 50 mg (N=6) | BIBF 1120 100 mg (N=8) | BIBF 1120 150 mg (N=24)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | BIBF 1120 50 mg (N=6) | BIBF 1120 100 mg (N=8) | BIBF 1120 150 mg (N=24)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Periproctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.